CLINICAL TRIAL: NCT06022211
Title: Post-COVID-19 Condition: Observational Study in Vietnam
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS 0268s POSTCOVIET
Record Dates: First submitted 2023-08-29; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Post COVID-19 Condition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — * 1 EDTA tube of 2 mL for complete blood count;
  * 1 heparinate tube of 2 mL for the biochemistry tests including glycaemia, transaminases, serum creatinine, CRP, ionogram (Na, K);
  * 1 EDTA tube of 2 mL for biobank (DBS and plasma).
  * 1 dry tube of 2 mL for HIV serology, HCV Ab, HBs Ag;
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this study is to estimate the prevalence of the post-COVID-19 condition in confirmed mild, moderate, and severe COVID-19 adult patients in Hai Phong, Vietnam.

DETAILED DESCRIPTION:
It is a cross-sectional study implemented in Hai Phong (Vietnam) by the Infectious and Tropical Diseases Department of Viet Tiep 2 hospital and the Department of Public Health of the Hai Phong University of Medicine and Pharmacy (HPMU).

The aim is to enroll moderate and severe COVID-19 patients from the 2 following provincial hospitals, Viet Tiep hospital and Kien An hospital, and mild COVID-19 patients from the community level in Hai Phong to assess the burden of post-COVID-19 condition in each patient group (mild, moderate or severe acute COVID-19).

835 participants are aimed to be interviewed through phone calls: 196 participants with mild disease, 289 participants with moderate disease, and 350 participants with severe disease. In case of suspected post-COVID-19 condition, the participant will be proposed to come to Viet Tiep 2 hospital for a study visit i) to confirm the post-COVID-19 condition, ii) to describe symptoms, iii) to evaluate the functional limitations related to the post-COVID-19 condition, and iv) to assess the determinants of the post-COVID-19 condition in patients with mild, moderate, and severe acute COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or more;
* With a history of documented COVID-19 as confirmed by either a positive SARS-CoV-2 RT-PCR or antigenic test, 3-12 months before inclusion;
* Hospitalised in Viet Tiep 2 hospital or Kien An hospital (tertiary care hospitals) with moderate or severe COVID-19 or registered in provincial CDC health system for mild COVID-19;
* Accepting to participate in the study;

Exclusion Criteria:

* Not able to understand or answer a quick phone questionnaire;
* Individuals who refuse or cannot come to Viet Tiep 2 hospital in case of the suspected post-COVID-19 condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients hospitalised in Viet Tiep 2 hospital or Kien An hospital for moderate or severe acute COVID-19 3 to 12 months before inclusion, or registered in the provincial CDC database for mild COVID-19 that occurred 3-12 months before inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 835 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the proportion of participants who present a post-COVID-19 condition in adult patients with confirmed mild, moderate, and severe COVID-19 in Hai Phong, Vietnam. | Day 0
  According to the WHO definition

SECONDARY OUTCOMES:
Type and frequency of symptoms of the post-COVID-19 condition. | Day 0
Functional limitations among participants with the post-COVID-19 condition. | Day 0
Factors related to occurrence of post-COVID-19 condition in adults after mild, moderate, and severe acute COVID-19. | Day 0